CLINICAL TRIAL: NCT01332357
Title: Use of Fluticasone Propionate/Salmeterol Combination Post Emergency Department Visit
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112606
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: fluticasone/propionate salmeterol combination; hospitalization; emergency department; asthma
MeSH Terms: conditions — Asthma; Emergencies | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Fluticasone propionate/salmeterol combination ED MD: Asthma subjects discharged from an institution after treatment for severe asthma exacerbation that receive fluticasone propionate/salmeterol combination from the ED physician
  Interventions: Drug: Fluticasone propionate/salmeterol combination ED MD
- Fluticasone propionate/salmeterol combination OP MD: Asthma subjects discharged from an institution after treatment for severe asthma exacerbation that receive fluticasone propionate/salmeterol combination from the OP physician
  Interventions: Drug: Fluticasone propionate/salmeterol combination OP MD

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol combination ED MD — Receipt of fluticasone propionate/salmeterol combination from the ED physician
  Groups: Fluticasone propionate/salmeterol combination ED MD
Drug: Fluticasone propionate/salmeterol combination OP MD — Receipt of fluticasone propionate/salmeterol combination from the OP physician
  Groups: Fluticasone propionate/salmeterol combination OP MD

SUMMARY:
The objective of this study is to compare readmission to the emergency department for asthma in asthma patients who receive treatment with fluticasone propionate and salmeterol oral inhaler after an initial emergency department visit using a retrospective observational cohort study design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with asthma as determined by ICD-9 codes and asthma drug use
* at least 12 years of age
* discharged from an initial Emergency Department visit within 12 months

Exclusion Criteria:

* Subjects with COPD or treatment for COPD

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study intends to identify subjects with asthma discharged from an emergency department that received fluticasone propionate/salmeterol from either an ED physician or from an outpatient physician
Sampling Method: Probability Sample
Enrollment: 6139 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not recruited for, nor enrolled in, this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Total Population: Adult and pediatric participants with persistent asthma were identified from commercially-insured and Medicaid health plan members with both medical and pharmacy benefits who had data in one of two healthcare claims databases.
Period: Overall Study
Arm/Group | Total Population
Started | 6139
Completed | 6139
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Population
Number analyzed (Participants) | 6139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.36 (17.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3392
  Male | 2747
Type of Index Event [Number; unit: visits] — The number of inpatient visits and emergency department visits that defined the index event are reported.
  visits
    Inpatient hospitalizations | 1331
    Emergency Department Visit | 4808
Charlson Comorbidity Index Scores [Mean (Standard Deviation); unit: scores on a scale] — The Charlson Comorbidity Index estimates 10-year mortality risk. Scores range from 0 - 37, with a lower score indicating a higher chance of survival.
  scores on a scale | 1.14 (0.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Asthma-related Event Occurring Between 1 and 6 Months Following the Index Event
Description: A subsequent asthma-related inpatient (IP) visit or emergency department (ED) visit were defined as visits within 6 months of the index event. The index event was defined as an asthma-related hospitalization or ED visit occuring between 2004 and 2008.
Time Frame: Data were collected during a 4-year period from January 1, 2004 to December 31, 2008.
Population: Adult and pediatric participants with persistent asthma were identified from commercially-insured and Medicaid health plan members with both medical and pharmacy benefits who had data in one of two healthcare claims databases.
Measure: Number; unit: participants
Arm/Group | Total Population
Number analyzed (Participants) | 6139
participants | 915
Statistical Analysis 1: Comparison: Total Population; Test type: Superiority or Other; p < 0.0001, Regression, Cox — The unadjusted risk of experiencing a recurrent event associated with not initiating a controller medication at index event discharge; Hazard Ratio (HR) = 1.96, 95% CI 2-sided [1.56 to 2.46]
Statistical Analysis 2: Comparison: Total Population; Test type: Superiority or Other; p < 0.0001, Regression, Cox — The adjusted risk of experiencing a recurrent event associated with not initiating a controller medication at index event discharge; Covariates included demographics, IP or ED index event, primary asthma diagnosis, Charlson score, and pre-index medication; Hazard Ratio (HR) = 1.79, 95% CI 2-sided [1.42 to 2.25]
Statistical Analysis 3: Comparison: Total Population; Test type: Superiority or Other; p < 0.0001, Regression, Cox — The risk of experiencing a recurrent event associated with not initiating a controller medication at index event discharge by time interaction; Evaluates the impact of each day treatment with a controller was delayed; Hazard Ratio (HR) = 1.008, 95% CI 2-sided [1.005 to 1.011]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical records and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Total Population
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.